CLINICAL TRIAL: NCT06521840
Title: Non-invasive Point-Of-Care Hemoglobin Testing In An Obstetric Population
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ethan Litman, Clinical Fellow in Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Other Study IDs: 2024P000128
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Masimo RAD 67 — This is an observational study of a non-invasive hemoglobin measurement device in a pregnant patient population. The current standard of care for anemia screening during pregnancy involves performing invasive venipuncture at two separate visits throughout the course of the pregnancy. The purpose of this research study is to compare the device performance with the gold standard hemoglobin measurement (venipuncture). The research team will use the Masimo Rad-67 handheld co-oximeter which has a reusable finger-tip sensor that enables spot-check monitoring measurements of both oxygen saturation and non-invasive hemoglobin measurement. At the time of a blood draw, the research team will place the pulse oximeter on the participant's finger. The devices requires 1-3 minutes for an accurate measurement. After the measurement is complete, the participant will be asked 2 questions on their satisfaction and comfortability with the device and 1 question regarding their skin tone.

SUMMARY:
Anemia is common during pregnancy due to increased metabolic rate and normal physiologic changes associated with pregnancy. Anemia during pregnancy has been associated with increased of adverse outcomes during delivery and the postpartum period. Currently, it is recommended to screen for anemia at three pre-specified points during routine prenatal care, typically 3 months apart. This screening method may miss patients who develop anemia between these intervals and lead to a delay in diagnosis and treatment.

MasimoTM has developed a non-invasive device that can detect anemia without a blood draw. This device has not been extensively studied in pregnant patients. The aim of this study is to determine the agreement in hemoglobin readings between the non-invasive device and the standard of care blood draws in pregnant patients.

DETAILED DESCRIPTION:
This is a prospective observational study of a non-invasive hemoglobin measurement device in a pregnant patient population. The device is FDA approved for use in adults, children, and neonates. The current standard of care for anemia screening during pregnancy involves performing invasive venipuncture at two separate visits throughout the course of the pregnancy. The purpose of this research study is to compare the device performance with the gold standard hemoglobin measurement (venipuncture) when patients receive routine hemoglobin measurement during the course of their prenatal care.

The research team will approach pregnant patients who are presenting for prenatal care at Beth Israel Deaconess Medical Center, including the Labor and Delivery Triage Unit. The research team also will approach patients during an antepartum or postpartum admission.

The research team will use the Masimo Rad-67 handheld co-oximeter which has a reusable finger-tip sensor that enables spot-check monitoring measurements of both oxygen saturation and non-invasive hemoglobin measurement. Study personnel will receive training on proper device use and cleaning by the local Masimo support team.

At the time of a blood draw, the research team will place the pulse oximeter on the participant's finger. The devices requires 1-3 minutes for an accurate measurement.

After the measurement is complete, the participant will be asked 2 questions on their satisfaction and comfortability with the device and 1 question regarding their skin tone using a validated skin tone scale.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or postpartum;
* Age ≥18 years old;
* Undergoing phlebotomy for clinical purpose

Exclusion Criteria:

- None

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant patients seeking prenatal care and pregnant patients admitted to the hospital for labor admission
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin (g /dL) Accuracy of Masimo RAD 67 | At time of phlebotomy
  Performance will be determined by calculating mean difference and repeatability analysis through the comparison of the hemoglobin values obtained from Masimo RAD67 to the hemoglobin values obtained from a reference phlebotomy sample collected at the same time.

SECONDARY OUTCOMES:
Hemoglobin (g /dL) Accuracy of Masimo RAD 67 stratified by skin tone | At time of phlebotomy
  Performance will be determined by calculating mean difference and repeatability analysis through the comparison of the hemoglobin values obtained from Masimo RAD67 to the hemoglobin values obtained from a reference phlebotomy sample collected at the same time stratified by skin color using a validated scale. Monk, Ellis. "The monk skin tone scale." (2019))
Hemoglobin (g /dL) Accuracy of Masimo RAD 67 stratified by gestational age | At time of phlebotomy
  Performance will be determined by calculating mean difference and repeatability analysis through the comparison of the hemoglobin values obtained from Masimo RAD67 to the hemoglobin values obtained from a reference phlebotomy sample collected at the same time stratified by gestational age.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No